CLINICAL TRIAL: NCT00198913
Title: Use of Modified Foods in the Dietary Treatment of Type II Diabetes Mellitus: Long Term Free Living Study
Brief Title: Long Term Free Living Study With Modified Foods and Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: American Diabetes Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADA2000-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2003-04

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Educational Status

INTERVENTIONS:
Behavioral: lower fat food supplied and education
Behavioral: gift cards for grocery foods and written education

SUMMARY:
Part 1 of this research demonstrated that type II diabetics are lacking in knowledge of how to best treat their illness with dietary controls. Most had little nutrition or diabetes knowledge. Part 2 demonstrated that providing a 40% reduction in fat intake across three meals versus all at one meal was more effective in glycemic control. Part 3 is designed to incorporate these findings into a long-term free living setting through education and behavior/dietary modification.

DETAILED DESCRIPTION:
Participants will be randomized into either the test group or the control group. Both groups will complete a one-week run-in period and then be followed over a 16 week period. This study will be conducted in two cohorts of 50 participants with 25 test participants and 25 control participants in each cohort.

Run-in Week - On the first day, participants will report to the laboratory for initial orientation to the study and methods. Baseline body measurements, height, weight and body composition analysis (using Bioelectrical Impendance), and a fasting blood sample, blood pressure and pulse will be taken. Participants will also complete additional study questionnaires and records. (Table 1 provides a summary of all measures at baseline and across the 16 week test period). Participants will also taste and rate various fat-replaced foods and complete a log of any changes in health over the next 3 days to determine palatability and tolerance of fat-replaced foods. Before trying foods, a survey will be administered to check for common food allergies. Finally, participants will be instructed to complete food diaries for 2 weekdays and 1 weekend day. Participants will return the food diaries and logs the following week. Participants who: 1) do not complete all parts of the run-in phase, 2) do not like and are not willing to eat at least 80% of the tested foods, or 3) have negative health effects following consumption of the foods will be dismissed from the study. No manipulations to participants' diets will occur during this phase.

16-Week Test Phase - During this phase, the test group will be given fat-replaced foods and instructed in a detailed diet plan to create a low-fat (<25% kcal from fat), weight maintenance diet providing optimal glycemic control. The test group will attend a 1h educational session (didactic and discussion) every 2wks. (Appendix 2 lists course topics.) Academic and professional staff will lead the sessions. Participants will be required to keep logs of certain behaviors and food records (2 weekdays and 1 weekend day over the 2wk period). Prior to the educational meetings, participants will submit data collection sheets (questionnaires and logs), be weighed and scheduled measures. Following the meeting, participants will be given fat-replaced foods for use over the next 2 weeks. Participants will be instructed to keep a log of usage of the provided foods, explicitly told that the foods are not for use by other members of their household and will be required to return all remaining or unused foods to the laboratory at the next meeting. In addition, at 8 weeks and 16 weeks, a blood sample, body composition, psychometrics, waist/hip measurements, blood pressure and pulse will be taken. The control group will receive vouchers for local supermarkets to offset the cost of the foods provided to the test group but will not be given actual food. This group will come to the laboratory every 2 weeks for identical data collection including blood draws but will not attend educational sessions. Instead, the control group will receive a newsletter every two weeks about the importance of a low-fat diet in the management of type II DM; however this newsletter will not give specific information about the use of fat-replaced foods in a low-fat diet. This newsletter will be sent to the test group as well.

Diet The test group diet plan will be designed to be a weight maintenance diet which derives no more than 25% kcal from fat (no more than 10% from saturated fat). A Registered Dietitian will design an individually tailored, 7d rotating suggested meal plan which includes the detailed use of fat-replaced foods according to the optimal strategy identified in Experiment 2. The individual prescriptions will be based upon the Mifflin-St.Joer equation and baseline intake obtained from the diet records from the run-in week.

ELIGIBILITY:
Inclusion Criteria:

type 2 diabetic, age 18 and over, informed consent,

Exclusion Criteria:

type 1 diabetic or non-diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-06; Study Completion 2003-02

PRIMARY OUTCOMES:
blood glucose control
weight

SECONDARY OUTCOMES:
body composition
psychometrics

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Lutherville, Maryland, United States